CLINICAL TRIAL: NCT00793013
Title: Primary Resuscitation Using Airway Pressure Release Ventilation Improves Recovery From Acute Lung Injury or Adult Respiratory Distress Syndrome and Reduces All Cause Mortality Compared to ARDS Net Low Tidal Volume-Cycled Ventilation.
Brief Title: Airway Pressure Release Ventilation (APRV) Compared to ARDSnet Ventilation
Acronym: PRESSURE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB approval lapsed.
Sponsor: University of Tennessee, Chattanooga (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123456789
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Acute Lung Injury; Adult Respiratory Distress Syndrome; Kidney Injury
Keywords: Acute Lung Injury; Adult Respiratory Distress Syndrome; Airway Pressure Release Ventilation; Acute Kidney Injury; Pressure Trial
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Acute Kidney Injury | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARDS Net Low Tidal Volume (Experimental)
  Interventions: Device: Volume-Cycled Assist-Control (AC) mode
- APRV Ventilation (Experimental)
  Interventions: Device: Airway Pressure Release Ventilation (APRV) mode

INTERVENTIONS:
Device: Volume-Cycled Assist-Control (AC) mode — 1. Patients ventilated with volume-cycled assist-control mode with PEEP and goal FIO2 < 40%
  2. Rate of mandatory time-cycled, pressure controlled breaths,initially at 12 per breaths/min
  3. Initial tidal volume set at 8mL/kg using predicted body weight (PBW) with a goal of 6mL/kg & setting positive end-expiratory pressure (PEEP) based on level of initial FiO2
  4. Inspiratory to Expiratory ratio set at 1:1 to 1:3
  5. If frequency of triggered breaths increased greater than 10 per min sedation will be increased. If needed,rate of mandatory breaths increased
  6. Mgmt of PEEP will be conducted as per the ARDSnet Protocol
  7. Oxygenation goal PaO2: PaO2-55-80 mm Hg O2 Sat: 88-95%
  8. Tidal volume and respiratory rate adjusted to the desired pH and plateau pressures per ARDSnet protocol
  Other Names: Controlled Mechanical Ventilation (CMV)
  Arms: ARDS Net Low Tidal Volume
Device: Airway Pressure Release Ventilation (APRV) mode — 1. Ventilation uses Drager Model X1
  2. Spontaneous breathing allowed throughout ventilatory cycle at 2 airway pressure levels
  3. Time periods for the high & low pressure levels can be set independently
  4. Duration of the lower pressure level will be adjusted to allow expiratory flow to decay to 75% of total volume
  5. Duration of higher pressure levels will be adjusted to produce 12 pressure shifts per min
  6. Spontaneous frequency will be targeted for 6 to 18 breaths/per min
  7. If spontaneous breathing is achieved,level of sedation will be decreased
  8. If spontaneous respirations are >20 breaths/min, sedation will be increased
  9. If spontaneous breathing frequency increased greater than 20/per min, sedation was increased and if needed the mechanical frequency increased
  Other Names: Controlled Mechanical Ventilation (CMV)
  Arms: APRV Ventilation

SUMMARY:
Traditional modes of ventilation have failed to improve patient survival. Subsequent observations that elevated airway pressures observed in traditional forms of ventilation resulted in barotrauma and extension of ALI lead to the evolution of low volume cycled ventilation as a potentially better ventilatory modality for ARDS. Recent multicenter trials by the NIH-ARDS network have confirmed that low volume ventilation increases the number of ventilatory free days and improves overall patient survival. While reducing mean airway pressure has reduced barotrauma and improved patient survival, it has impaired attempts to improve alveolar recruitment. Alveolar recruitment is important as it improves V/Q mismatch, allows reduction in FIO2 earlier, and decreases the risk of oxygen toxicity. Airway pressure release ventilation (APRV) is a novel ventilatory modality that utilizes controlled positive airway pressure to maximize alveolar recruitment while minimizing barotrauma. In APRV, tidal ventilation occurs between the increase in lung volumes established by the application of CPAP and the relaxation of lung tissue following pressure release. Preliminary studies have suggested that APRV recruits collapsed alveoli and improves oxygenation through a restoration of pulmonary mechanics, but there are no studies indicating the potential overall benefit of APRV in recovery form ALI/ADRS.

DETAILED DESCRIPTION:
Low volume ventilation may increase number of ventilatory free days and may improve overall patient survival. While reducing mean airway pressure has reduced barotrauma and improved patient survival, it has impaired attempts to improve alveolar recruitment. Alveolar recruitment is important as it improves V/Q mismatch, allows reduction in FIO2 earlier, and decreases the risk of oxygen toxicity. Airway pressure release ventilation (APRV) is a novel ventilatory modality that utilizes controlled positive airway pressure to maximize alveolar recruitment while minimizing barotrauma. In APRV, tidal ventilation occurs between the increase in lung volumes established by the application of CPAP and the relaxation of lung tissue following pressure release. Preliminary studies have suggested that APRV recruits collapsed alveoli and improves oxygenation through a restoration of pulmonary mechanics, but there are no studies indicating the potential overall benefit of APRV in recovery form ALI/ADRS.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Internal Medicine service at the Baroness Erlanger Hospital of the University of Tennessee College of Medicine with hypoxia (O2 saturation < 93%) and pulmonary distress, will be screened for study participation.
* Patients displaying all the following clinical criteria: acute onset of respiratory failure; hypoxia defined as a PaO2/FiO2 ratio of < 300 Torr; pulmonary capillary wedge pressure less or equal than 18 mm Hg, and/or no clinical evidence of left sided heart failure; and chest x-ray with diffuse bilateral pulmonary infiltrates.

Exclusion Criteria:

* Patients receiving conventional volume ventilation with or without PEEP for > 6 hours prior to study enrollment
* Patient's family or surrogate unwilling to give informed consent
* Patients requiring sedation or paralysis for effective ventilation
* Patients known pulmonary embolus within 72 hours of study enrollment
* Patients with close head injuries or evidence of increased intracranial pressure
* Patients with burns over 30% of total body surface area
* Pulmonary capillary wedge pressure greater than 18 mm Hg
* CVP > 15 cm H2O
* Patients with B type Naturetic peptide levels > 1000
* Patients with prior history of dilated cardiomyopathy with EF < 25%
* Patients receiving chronic outpatient peritoneal or hemodialysis
* Patients with severe liver disease (as defined by Child-Pugh class C)
* AIDS patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 28 days or prior to hospital discharge

SECONDARY OUTCOMES:
Number of ventilator-free days | 28 days or prior to hospital discarge
Length of ICU stay and /or Total hospital days | 28 days or prior to hospital discharge
To determine the effects of APRV ventilation versus ARDS net low volume-cycle ventilation on the incidence of of AKI | 28 days or prior to hospital discharge
To determine the effects of APRV ventilation versus ARDS net low volume-cycle ventilation on the NGAL, KIM-1, and IL-18 urine biomarkers for AKI | 28 days or prior to hospital discharge
To determine the effects of APRV ventilation versus ARDS net low volume-cycle ventilation in maintaining hourly urine output > 0.5 mls/kg/hr | 28 days or prior to hospital discharge
Will determine urinary aquaporin-2 levels in patients randomized to APRV ventilation versus ARDS net low volume-cycle ventilation | 28 days or prior to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: James A Tumlin, MD, Principal Investigator — University of Tennessee
Locations (1):
- James A. Tumlin, MD, Chattanooga, Tennessee, United States